CLINICAL TRIAL: NCT04759391
Title: Effects of Digital Pelvic Floor Muscle Training and Lifestyle Recommendations in Patients With Multiple Sclerosis Having Lower Urinary Tract Symptoms
Brief Title: Effects of Digital Pelvic Floor Muscle Training in Patients With Multiple Sclerosis Having Lower Urinary Tract Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, associate professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/02/15
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Multiple Sclerosis; Pelvic Floor Muscle Training
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups (control and exercise) for treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Lifestyle recommendations as well as digital pelvic floor muscle training to the exercise group
  Interventions: Other: Exercise; Other: Lifestyle recommendations
- Control group (Active Comparator): Lifestyle recommendations will be given to the control group
  Interventions: Other: Lifestyle recommendations

INTERVENTIONS:
Other: Exercise — Pelvic floor muscle training program planned under the supervision of a physiotherapist was applied and followed to the exercise group, using the digital application.
  Arms: Exercise group
Other: Lifestyle recommendations — Information was given within the scope of lifestyle recommendations (fluid intake, diet, constipation, weight control, smoking related to lower urinary system symptoms

SUMMARY:
The aim of this study was to investigate the effects of digital pelvic floor muscle training and lifestyle recommendations in patients with Multiple Sclerosis having lower urinary tract symptoms.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune, neurodegenerative disease of the central nervous system. Lower urinary tract symptoms (LUTS) are very common in MS. Pelvic floor muscle training (PFMT) is one of the first-line choices for the conservative treatment of LUTS.

According to our knowledge, no study has investigated the effects of digital pelvic floor muscle training and lifestyle recommendations in MS having LUTS, yet.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of MS and having at least two of the lower urinary symptoms
* Not having an attack in the last 1 month,
* No change in medical treatment in the last 3 months
* "Expanded disability status scale-EDSS" score is less than 6.5
* Not having any cognitive problems that would hinder cooperation and understanding
* Those who use digital devices such as computers, laptops, smartphones and tablets
* Volunteering to participate in the study

Exclusion Criteria:

* Pregnancy status
* Active urinary tract infection
* Another neurological disease that can cause incontinence
* A history of malignancy
* Prostate surgery
* Those with missing evaluation parameters
* Those who do not regularly participate in treatment programs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Incontinence symtoms | change from baseline at 8 weeks
  Urinary incontinence symptoms will be evaluated with The International Consultation of Incontinence Questionnaire - Short Form
Overactive bladder symptoms | change from baseline at 8 weeks
  Overactive bladder symptoms will be evaluated with Overactive Bladder Questionnaire-Version8

SECONDARY OUTCOMES:
bladder functions | change from baseline at 8 weeks
  bladder functions will be evaluated with voiding diary
Quality of life level | change from baseline at 8 weeks
  Quality of life will be evaluated with King's Health Questionnaire
subjective perception of improvement | after treatment (8th week)
  subjective perception of improvement will be evaluated with a 4-item Likert-type scale
patient satisfaction | after treatment (8th week)
  patient satisfaction will be evaluated with a 5-item Likert-type scale

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No